CLINICAL TRIAL: NCT06950996
Title: An in Silico External Clinical Validation of AI Solutions for Cancer Management in the CHAIMELEON Project. Applied to 4 Target Types of Cancer (Lung, Breast, Prostate and Colorectal), Collected Through the Routine Delivery of Health Care With no Enrolment Conditinos (Real World Data).
Brief Title: A Clinical Evaluation of AI Solutions Developed in the CHAIMELEON Project for Cancer: Prostate, Lung, Breast, Colon and Rectum
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: University of Pisa (Other); University Hospital Rijeka (Other); University of Messina (Other); Istanbul Medipol University Hospital (Other); Centro Hospitalar do Porto (Other); Hospitales Universitarios Virgen del Rocío (Other); IRCCS Policlinico S. Donato (Other); National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other); Charite University, Berlin, Germany (Other); Osakidetza (Other); Le Collège des Enseignants de Radiologie de France (Other)
Responsible Party: Sponsor
Other Study IDs: CHAIMELEON insilico validation; 952172 (Other Grant/Funding Number: European Union's Horizon 2020)
Record Dates: First submitted 2025-04-11; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Lung Cancer, Non-Small Cell; Colon Cancer; Rectum Cancer; Prostate Cancer
Keywords: Clinical validation; AI model solutions; experimental dedicated-platform
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms; Prostatic Neoplasms | interventions — Risk; Life Expectancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Evaluation with Medical expertise only: Evaluation of different medical images of people with 5 types of cancer using their own expertise.
  Interventions: Other: Risk in prostate cancer; Other: Life expectancy in lung cancer; Other: Histological subtype; Other: Staging of colon cancer; Other: invasion in rectum cancer
- Group 2: Evaluation with the support of AI solutions: Evaluation of different medical images of people with 5 types of cancer guided by the AI solutions developed.
  Interventions: Other: Risk in prostate cancer; Other: Life expectancy in lung cancer; Other: Histological subtype; Other: Staging of colon cancer; Other: invasion in rectum cancer

INTERVENTIONS:
Other: Risk in prostate cancer — the prediction involves the classification of the prostate cancer according to the level of prostatic antigen (PSA), the biopsy classification of the aggressiveness of the tumour, and also the localisation of the tumour
Other: Life expectancy in lung cancer — Clinicians will evaluate life expectancy in lung cancer using CTs, together with some clinical information.
Other: Histological subtype — An assessment by pathology of the subtype of breast tumour
Other: Staging of colon cancer — classify size, lymph node involvement and possibility of metastasis in medical images (computerized tomosynthesis) of thorax and pelvis region
Other: invasion in rectum cancer — assess whether vascular extramural o mesorectal fascia has been invaded in the tumour using magnetic resonance medical images taken at diagnosis in the pelvic region

SUMMARY:
The goal of this observational study is to see how useful an experimental viewer and AI solutions are for clinicians in their daily work. The investigators want to find out if the AI helps clinicians interpret medical images for different types of cancer.

The AI solutions aim to:

* Classify whether prostate cancer is low or high risk
* Classify the histological subtype in breast cancer
* Estimate the life expectancy of patients with lung cancer
* Determine the size of colon cancer, lymph node involvement and the possibility of metastasis..
* Assess the invasion of sorrounding tissues in the case of rectum cancer. The study will involve clinicians from various centres who will review a set of cases not previously analysed by the AI. Clinicians will do this in two phases: first using only their own expertise and then with the help of the AI solutions.

The technical team want to see if the AI solutions assist clinicians and could become useful in the everyday clinical practice. Clinicians will complete a survey to share their feedback on the usability of the platform and how helpful the AI solutions are.

DETAILED DESCRIPTION:
In order to conduct a robust clinical validation, the investigators have designed a study on the required sample size. The study is design to evaluate the role of an AI-assisted tool as a support for improving the daily clinical work. The investigators used an online website (https://statulator.com/SampleSize/ss2PP.html) for the calculation and use the "paired binary proportions" option. Using the case of prostate cancer, the investigators want to compare the probability of correct risk classification in prostate cancer by clinicians alone and/or guided by AI. The study will have a significance (α) = 0.05; power (β) = 80%; the analysis will be "two sided" and with equal group sizes.

An 10% improvement in cancer risk classification was observed when clinicians had access to an AI tool solution (Yilmaz et al.,). In addition, the authors reported that expert readers had an accuracy rate of 81% compared to 69% for novice readers when determining the Gleason score of lesions (a medical term used in pathology to classify the aggressiveness of cells in a tumour). The authors also assumed an 80% correlation between paired observations.

As a result, at least 60 new cases would be needed to evaluate the performance of the AI tool.

ELIGIBILITY:
Inclusion Criteria:

* patients with an histological confirmation of cancer diagnosis (prostate, lung, breast, colon or rectum)
* availability of radiological images (MR for prostate and rectum, CT for lung and colon or mammographys for breast).
* enough follow up (12 months for prostate, breast and rectum), 18 months for lung, and 24 months for colon.

Exclusion Criteria:

* patients with incomplete or low quality data (radiological, pathological or uncomplete clinical data necessary for the ground truth)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a cancer diagnosis of prostate, breast, lung and colorectal from the University and politechnic Hospital la Fe, Valencia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Usability of experimental viewer with AI tools | 5 months
  Usability of the platform was assessed at the end of each of the two study phases: a standard clinical phase (without artificial intelligence assistance) and a second phase assisted by AI models. Participants evaluated their experience using a 5-point Likert scale, where 1 indicated "strongly disagree" and 5 indicated "strongly agree," in response to statements regarding ease of use, interface clarity, system efficiency, overall satisfaction, and other aspects related to user interaction with the platform.
  This assessment enabled a comparison of user perceptions of the viewer's usability under both conventional clinical conditions and AI-assisted conditions. Higher scores reflect a better user experience.
Utility of experimental medical images viewer | 5 months
  The utility of the experimental viewer was assessed by comparing clinicians' diagnostic accuracy and time spent when using the system alone versus with AI assistance. Higher accuracy and reduced interpretation time were considered indicators of greater utility. The goal was to determine whether the viewer enhances clinical decision-making, streamlines workflows, and supports better patient care.
  Additional data such as clinician gender, specialty, and experience were collected to enable subgroup analyses. Statistical evaluations included confusion matrices to assess diagnostic performance, and Sankey flow diagrams to visualize changes in decision-making between unaided and AI-assisted phases. These tools provided a comprehensive understanding of the viewer's practical benefit in real clinical scenarios.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico la Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz EC, Turkbey B. The added value of a deep learning-based computer-aided detection system on prostate cancer detection among readers with varying level of multiparametric MRI expertise. Chin Clin Oncol. 2022 Dec;11(6):42. doi: 10.21037/cco-22-104. Epub 2022 Nov 15. No abstract available. PMID 36408543
- See also: Accelerating the lab to market transition of AI tools for cancer management is an European project that contemplates the evaluation of the in silico clinical validation — https://chaimeleon.eu